CLINICAL TRIAL: NCT03148457
Title: Early Versus Late Initiation of Direct Oral Anticoagulants in Post-ischaemic Stroke Patients With Atrial fibrillatioN (ELAN): an International, Multicentre, Randomised-controlled, Two-arm, Assessor-blinded Trial
Acronym: ELAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00588
Record Dates: First submitted 2017-04-07; First posted 2017-05-11 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Ischaemic Stroke
Keywords: Stroke; Direct oral anticoagulation; Apixaban; Dabigatran; Rivaroxaban; Edoxaban; Therapy initiation; Major bleeding; Atrial fibrillation
MeSH Terms: conditions — Ischemic Stroke; Stroke; Atrial Fibrillation | interventions — Rivaroxaban; Dabigatran; apixaban; edoxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early treatment (Experimental): Early treatment of patients with ischaemic stroke related to atrial fibrillation (AF) with direct oral anticoagulations (DOACs).
  Interventions: Drug: Early treatment with Rivaroxaban (Xarelto®), Dabigatran (Pradaxa®), Apixaban (Eliquis®) or Edoxaban (Lixiana®)
- Late treatment (Other): Treatment with direct oral anticoagulations (DOACs) according the current standard practice in patients with acute ischemic stroke related to atrial fibrillation (AF).
  Interventions: Drug: Late treatment with Rivaroxaban (Xarelto®), Dabigatran (Pradaxa®), Apixaban (Eliquis®) or Edoxaban (Lixiana®)

INTERVENTIONS:
Drug: Early treatment with Rivaroxaban (Xarelto®), Dabigatran (Pradaxa®), Apixaban (Eliquis®) or Edoxaban (Lixiana®) — Early treatment will be started within 48 hours after symptom onset (minor and moderate ischaemic stroke) or at day 6 + 1 day after symptom onset (major ischaemic stroke)
  Arms: Early treatment
Drug: Late treatment with Rivaroxaban (Xarelto®), Dabigatran (Pradaxa®), Apixaban (Eliquis®) or Edoxaban (Lixiana®) — Patients in the control arm will receive late treatment as per current recommendations (i.e. minor ischaemic stroke after day 3 + 1 day, moderate ischaemic stroke after day 6 + 1 day and major ischaemic stroke after day 12 + 2 day).
  Arms: Late treatment

SUMMARY:
When to start anticoagulation in patients with an acute ischaemic stroke and atrial fibrillation (AF) is a relevant unanswered question in clinical practice. Direct oral anticoagulants (DOACs) are highly effective for secondary stroke prevention in these patients, but DOACs were never initiated <7 days after stroke onset in recent trials. The ELAN trial will determine the net benefit of early versus late initiation of DOACs in patients with acute ischaemic stroke related to AF.

The main objective is to estimate the net benefit of early versus late initiation of DOACs in patients with acute ischaemic stroke related to AF.

The secondary objectives are to assess all vascular events and all-cause mortality after early initiation of DOACs in patients with acute ischaemic stroke related to AF compared to late initiation.

DETAILED DESCRIPTION:
Background Atrial fibrillation (AF) is the most common cardiac arrhythmia increasing the risk of stroke and systemic thromboembolism and thus mortality and morbidity. Anticoagulation therapy, such as with vitamin K antagonists effectively prevents strokes in patients with AF, however, increases bleeding complications leading to symptomatic intracerebral haemorrhage. Direct oral anticoagulants (DOACs) are at least as effective as vitamin K antagonists in preventing recurrent strokes, but with lower rates of symptomatic intracerebral haemorrhage. Therefore, these new agents are potentially ideal drugs to treat patients with ischaemic stroke related to AF. However, in previous trials comparing DOACs with vitamin K antagonists, therapy was initiated later than 7-14 days after onset of ischaemic stroke. Whether, earlier initiation of DOACs may prevent recurrent stroke without increasing the risk of symptomatic intracerebral haemorrhage remains to be determined.

Objectives The main objective is to estimate the net benefit of early versus late initiation of DOACs in patients with acute ischaemic stroke related to AF.

The secondary objectives are to assess all vascular events and all-cause mortality after early initiation of DOACs in patients with acute ischaemic stroke related to AF compared to late initiation.

Methods All patients of 18 years or older with an acute ischaemic stroke related to AF should be screened for this trial.

Patients in the experimental arm (early treatment) and the control arm (late treatment) will receive direct oral anticoagulants for prevention of stroke and systemic embolism in patients with AF. Depending on the size of the infarction, early treatment will be started within 48 hours after symptom onset (minor and moderate ischaemic stroke) or at day 6 + 1 day after symptom onset (major ischaemic stroke). Patients in the control arm will receive late treatment as per current recommendations (i.e. minor ischaemic stroke after day 3 + 1 day, moderate ischaemic stroke after day 6 + 1 day and major ischaemic stroke after day 12 + 2 day).

The primary outcome is a composite of major bleeding, recurrent ischaemic stroke, systemic embolism and/or vascular death at 30 ± 3 days after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to country specific details
* Age: ≥18 years
* Acute ischemic stroke, either confirmed by MRI or CT scan (tissue based definition) or by sudden focal neurological deficit of presumed ischaemic origin that persisted beyond 24 hours and otherwise normal non-contrast CT scan. Please note: prior intravenous or endovascular treatment is allowed.
* Permanent, persistent, or paroxysmal spontaneous AF previously known or diagnosed during the index hospitalization
* Agreement of treating physician to prescribe DOACs

Exclusion Criteria:

* Atrial fibrillation due to reversible causes (e.g. thyrotoxicosis, pericarditis, recent surgery, myocardial infarct)
* Valvular disease requiring surgery
* Mechanical heart valve(s)
* Moderate or severe mitral stenosis. Please note that other valvular diseases and biological valves are eligible
* AF and conditions other than AF that require anticoagulation, including therapeutical dose of low-molecular-weight heparin or heparin. Please note: infratherapeutic anticoagulation at ischaemic stroke onset defined as follows is not an exclusion criteria:

  * Vitamine K antagonist: International Normalized Ratio (INR) <1.7
  * Anti-IIa: thrombin time <80 seconds and/or anti-IIa <50 ng/ml
  * Anti-Xa: anti-Xa <50 ng/ml
* Subject who is contraindicated to DOACs
* Female who is pregnant or lactating or has a positive pregnancy test at time of admission
* Patients with serious bleeding in the last 6 months or is at high risk of bleeding (e.g. active peptic ulcer disease, platelet count < 100'000/mm3 or haemoglobin < 10 g/dl or INR ≥ 1.7, documented haemorrhagic tendencies or blood dyscrasias)
* Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day)
* Severe comorbid condition with life expectancy < 6 months
* Severe or moderate renal insufficiency as defined by creatinine clearance < 50 ml/min
* Subject who requires haemodialysis or peritoneal dialysis
* Subject with aortic dissection
* Current participation in another investigational trial
* Dual antiplatelet therapy at baseline or strong likelihood to be treated with dual antiplatelet therapy during the course of the trial
* CT or MRI evidence of haemorrhage classified as PH1 (defined as parenchymal haemorrhage = blood clots in <30% of the infarcted area without or with slight space-occupying effect) and PH2 (defined as blood clots in >30% of the infarcted area with a substantial space-occupying effect) independently of clinical deterioration. Please note that HI1 (defined as haemorrhagic infarct = small petechiae along the margins of the infarct) and HI2 (defined as confluent petechiae within the infarcted area but no space occupying effect) are acceptable if not associated with clinical deterioration and if the treating physician feels comfortable to treat patients with DOACs.
* CT or MRI evidence of mass effect or intra-cranial tumour (except small meningioma)
* CT or MRI evidence of cerebral vasculitis
* Endocarditis
* Evidence of severe cerebral amyloid angiopathy if MRI scan performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2013 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Composite of major bleeding, recurrent ischaemic stroke, systemic embolism and/or vascular death | 30 ± 3 days after randomisation

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 30 days, 90 days after randomisation
Major bleeding | 30 days, 90 days after randomisation
Non-major bleeding | 30 days, 90 days after randomisation
Recurrence of stroke | 30 days, 90 days after randomisation
Systemic embolism | 30 days, 90 days after randomisation
Vascular death | 30 days, 90 days after randomisation
All-cause mortality | 90 days after randomisation
Myocardial infarction | 90 days after randomisation
Major cardiovascular events defined as composite of stroke, myocardial infarct, heart failure or cardiovascular death | 90 days after randomisation
Silent brain lesions | 90 days after randomisation
  If CT/MRI is performed in clinical routine
Favourable outcome defined as mRS ≤ 2 and shift analysis adjusted to premorbid mRS | 90 days after randomisation
NIHSS | 90 days after randomisation
Transient ischemic attack | 30 days, 90 days after randomisation
Undetermined stroke | 30 days, 90 days after randomisation
Compliance | 30 days after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, Prof. MD, Principal Investigator — Dept. of Neurology, Inselspital Bern
Locations (98):
- Austria (7):
  - Krankenhaus der Barmherzigen Brüder Eisenstadt, Eisenstadt
  - Medizinische Universität Graz, Graz
  - Kepler Universitätsklinikum, Klinik für Neurologie 1, Linz
  - Kepler Universitätsklinikum, Klinik für Neurologie 2, Linz
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Universitätsklinikum Tulln, Tulln
  - Medizinische Universität Wien, Vienna
- Belgium (8):
  - Onze-Lieve-Vrouw Ziekenhuis VZW, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - University Hospital Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC - Saint Joseph, Liège
  - Cliniques de l'Europe - Site Ste-Elisabeth, Uccle
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Siun sote - North Karelia social and health services, Joensuu
- Germany (12):
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Vivantes Klinikum Neukölln, Berlin
  - St. Josef-Hospital Bochum, Bochum
  - Klinik und Poliklinik für Neurologie Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Neurologische Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Mannheim University Hospital, Mannheim
  - Klinikum der Universität München, München
  - Universitäsklinikum Tübingen, Tübingen
- Dept. of Medicine, University of Thessaly, Larissa, Thessaly, Greece
- India (7):
  - Lalitha Super Speciality Hospitals, Kothapeta, Guntur
  - Narayana Hrudayalaya Bangalore, Bengaluru, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Government Medical College Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Trivandrum, Kerala
  - All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Christian Medical College & Hospital, Ludhiana, Punjab
- Ireland (6):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Waterford, Waterford
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Centre, Ramat Gan
- Italy (2):
  - Ospedale Santa Maria della Misericordia, Perugia
  - Umberto Policlinico di Roma, Rome
- Japan (6):
  - Kansai Medical University, Hirakata
  - St. Marianna Medical University Hospital, Kawasaki
  - Kumamoto University, Kumamoto
  - National Cerebral and Cardiovascular Center, Osaka
  - Jichi Medical University, Tochigi
  - The Jikei University Hospital, Tokyo
- Norway (4):
  - Ålesund sjukehus, Ålesund
  - Vestre Viken Health Trust - Drammen Hospital, Drammen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Ullevål, Oslo
- Portugal (3):
  - Coimbra University Hospital, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Hospital de Egas Moniz, Lisbon
- Slovakia (2):
  - Košice Medical University, Košice
  - Fakultná Nemocnica Trnava, Trnava
- Switzerland (18):
  - Dept. of Neurology, Kantonsspital Aarau, Aarau, Canton of Aargau
  - Dept. of Neurology, Universitätsspital Basel, Basel, Canton of Basel-City
  - Dept. of Neurology, Universitätsspital Lausanne, Lausanne, Canton of Vaud
  - Dept. of Neurology, Hôpital de Zone de Nyon, Nyon, Canton of Vaud
  - Dept. of Neurology, Kantonsspital Chur, Chur, Kanton Graubünden
  - Dept. of Neurology, Kantonsspital Sion, Sion, Valais
  - Kantonsspital Baden, Baden
  - Dept. of Neurology, Bern University Hospital, Bern
  - Dept. of Neurology, Kantonsspital Fribourg, Fribourg
  - Dept. of Neurology, Universitätsspital Genf, Geneva
  - Dept. of Neurology, Kantonsspital Luzern, Lucerne
  - Ospedale Regionale di Lugano (EOC), Lugano
  - Kantonsspital Münsterlingen, Münsterlingen
  - Hôpital neuchâtelois, Neuchâtel
  - Dept. of Neurology, Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden Zürich, Zurich
  - Dept. of Neurology, Universitätsspital Zürich, Zurich
- United Kingdom (17):
  - St George's University Hospitals NHS Foundation Trust, Tooting, London
  - University Hospital Monklands, Airdrie
  - Royal United Hospitals Bath, Bath
  - Southmead Hospital Bristol, Bristol
  - Countess of Chester Hospital, Chester
  - Ninewells Hospital, Dundee
  - University Hospital of North Durham, Durham
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Wirral University Teaching Hospital, Metropolitan Borough of Wirral
  - The James Cook University Hospital, Middlesbrough
  - Morriston Hospital, Morriston
  - Perth Royal Infirmary, Perth
  - Glan Clwyd Hospital, Rhyl
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Weston General Hospital, Weston-super-Mare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polymeris AA, Rossel JB, Koga M, Strbian D, Vedamurthy A, Krishnan M, Branca M, Meinel T, Kristoffersen ES, Yoshimoto T, Tanaka K, Kunieda T, Yakushiji Y, Vehoff J, Matsuzono K, Slade P, Demeestere J, Salerno A, Caracciolo NG, Hemelsoet D, Engelter ST, Auer E, Horvath T, Seiffge DJ, Goeldlin M, Dawson J, Fischer U. Once- versus twice-daily direct oral anticoagulants after ischemic stroke in atrial fibrillation - A post-hoc analysis of the ELAN trial. Eur Stroke J. 2026 Jan 1;11(1):23969873251360974. doi: 10.1093/esj/23969873251360974. PMID 41614485
- [Derived] Polymeris AA, Rossel JB, Koga M, Strbian D, Vedamurthy A, Krishnan M, Branca M, Meinel T, Kristoffersen ES, Yoshimoto T, Tanaka K, Kunieda T, Yakushiji Y, Vehoff J, Matsuzono K, Slade P, Demeestere J, Salerno A, Caracciolo NG, Hemelsoet D, Engelter ST, Auer E, Horvath T, Seiffge DJ, Goeldlin M, Dawson J, Fischer U; ELAN Investigators. Once- versus twice-daily direct oral anticoagulants after ischemic stroke in atrial fibrillation - A post-hoc analysis of the ELAN trial. Eur Stroke J. 2025 Aug 11:23969873251360974. doi: 10.1177/23969873251360974. Online ahead of print. PMID 40785636
- [Derived] Wouters A, Demeestere J, Rossel JB, Devroye A, Desfontaines P, Vanacker P, Hemelsoet D, Yperzeele L, Rutgers MP, Peeters A, Vynckier J, Yoshimoto T, Tanaka K, Vehoff J, Matsuzono K, Kulyk C, Sibolt G, Slade P, Salerno A, Kunieda T, Hakim A, Rohner R, Abend S, Goeldlin M, Dawson J, Fischer U, Lemmens R; ELAN Investigators. Prior Reperfusion Strategy Does Not Modify Outcome in Early Versus Late Start of Anticoagulants in Patients With Ischemic Stroke: Prespecified Subanalysis of the Randomized Controlled ELAN Trial. Stroke. 2025 Aug;56(8):2000-2008. doi: 10.1161/STROKEAHA.125.050646. Epub 2025 May 22. PMID 40402090
- [Derived] Kneihsl M, Hakim A, Goeldlin MB, Branca M, Fenzl S, Abend S, Gattringer T, Enzinger C, Dawson J, Gesierich B, Kopczak A, Hack RJ, Cerfontaine MN, Rutten JW, Lesnik Oberstein SAJ, Pasi M, Fischer U, Duering M, Meinel TR. Topographic Localization of Chronic Cerebellar Ischemic Lesions: Implications for Underlying Cause. Stroke. 2025 Jul;56(7):1823-1831. doi: 10.1161/STROKEAHA.124.049337. Epub 2025 Apr 3. PMID 40177749
- [Derived] Polymeris AA, Branca M, Sylaja PN, Sandset EC, de Sousa DA, Thomalla G, Paciaroni M, Gattringer T, Strbian D, Trelle S, Michel P, Nedeltchev K, Bonati LH, Ntaios G, Koga M, Gdovinova Z, Lemmens R, Bornstein NM, Kelly P, Goeldlin MB, Abend S, Selim M, Katan M, Horvath T, Dawson J, Fischer U; ELAN Investigators. Net Benefit of Early Anticoagulation for Stroke With Atrial Fibrillation: Post Hoc Analysis of the ELAN Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2456307. doi: 10.1001/jamanetworkopen.2024.56307. PMID 39874037
- [Derived] Kneihsl M, Hakim A, Goeldlin MB, Meinel TR, Branca M, Rohner R, Fenzl S, Abend S, Shim GC, Gumbinger C, Zhang L, Kristoffersen ES, Desfontaines P, Vanacker P, Alonso A, Poli S, Nunes AP, Caracciolo NG, Gattringer T, Kahles T, Giudici D, Demeestere J, Dawson J, Fischer U; ELAN investigators. Early vs Late Anticoagulation After Ischemic Stroke in Patients With Atrial Fibrillation and Covert Brain Infarcts. Neurology. 2025 Jan 14;104(1):e210157. doi: 10.1212/WNL.0000000000210157. Epub 2024 Dec 19. PMID 39700448
- [Derived] Goeldlin MB, Hakim A, Branca M, Abend S, Kneihsl M, Valenzuela Pinilla W, Fenzl S, Rezny-Kasprzak B, Rohner R, Strbian D, Paciaroni M, Thomalla G, Michel P, Nedeltchev K, Gattringer T, Sandset EC, Bonati L, Aguiar de Sousa D, Sylaja PN, Ntaios G, Koga M, Gdovinova Z, Lemmens R, Bornstein NM, Kelly P, Katan M, Horvath T, Dawson J, Fischer U; ELAN Investigators. Early vs Late Anticoagulation in Minor, Moderate, and Major Ischemic Stroke With Atrial Fibrillation: Post Hoc Analysis of the ELAN Randomized Clinical Trial. JAMA Neurol. 2024 Jul 1;81(7):693-702. doi: 10.1001/jamaneurol.2024.1450. PMID 38805207
- [Derived] Rohner R, Kneihsl M, Goeldlin MB, Hakim A, Branca M, Abend S, Valenzuela Pinilla W, Fenzl S, Rezny-Kasprzak B, Strbian D, Trelle S, Paciaroni M, Thomalla G, Michel P, Nedeltchev K, Gattringer T, Sandset EC, Bonati L, Aguiar de Sousa D, Sylaja PN, Ntaios G, Koga M, Gdovinova Z, Lemmens R, Bornstein NM, Kelly P, Katan M, Horvath T, Dawson J, Fischer U; ELAN Investigators. Early Versus Late Initiation of Direct Oral Anticoagulants After Ischemic Stroke in People With Atrial Fibrillation and Hemorrhagic Transformation: Prespecified Subanalysis of the Randomized Controlled ELAN Trial. Circulation. 2024 Jul 2;150(1):19-29. doi: 10.1161/CIRCULATIONAHA.124.069324. Epub 2024 May 16. PMID 38753452
- [Derived] Fischer U, Koga M, Strbian D, Branca M, Abend S, Trelle S, Paciaroni M, Thomalla G, Michel P, Nedeltchev K, Bonati LH, Ntaios G, Gattringer T, Sandset EC, Kelly P, Lemmens R, Sylaja PN, Aguiar de Sousa D, Bornstein NM, Gdovinova Z, Yoshimoto T, Tiainen M, Thomas H, Krishnan M, Shim GC, Gumbinger C, Vehoff J, Zhang L, Matsuzono K, Kristoffersen E, Desfontaines P, Vanacker P, Alonso A, Yakushiji Y, Kulyk C, Hemelsoet D, Poli S, Paiva Nunes A, Caracciolo N, Slade P, Demeestere J, Salerno A, Kneihsl M, Kahles T, Giudici D, Tanaka K, Raty S, Hidalgo R, Werring DJ, Goldlin M, Arnold M, Ferrari C, Beyeler S, Fung C, Weder BJ, Tatlisumak T, Fenzl S, Rezny-Kasprzak B, Hakim A, Salanti G, Bassetti C, Gralla J, Seiffge DJ, Horvath T, Dawson J; ELAN Investigators. Early versus Later Anticoagulation for Stroke with Atrial Fibrillation. N Engl J Med. 2023 Jun 29;388(26):2411-2421. doi: 10.1056/NEJMoa2303048. Epub 2023 May 24. PMID 37222476